CLINICAL TRIAL: NCT04958213
Title: Isokinetic Evaluation of the Efficacy of Dextrose Prolotherapy Treatment in Women With Knee Osteoarthritis.
Brief Title: The Effect of Dextrose Prolotherapy on Isokinetic Power in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Kamil Mursit Yildiz, Research assistant, Mustafa Kemal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MustafaKU-KOA-Prolo
Record Dates: First submitted 2021-06-30; First posted 2021-07-12 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Knee Osteoarthritis; Dextrose Prolotherapy Injection; Physical Therapy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional physical therapy (Other): Conventional physical therapy (Hotpack, TENS and Ultrasound) and home exercise program (isometric and isotonic exercises) will be applied to this group for 4 weeks (20 sessions).
  Interventions: Combination Product: conventional physical therapy
- Dextrose prolotherapy treatment (Active Comparator): This group will be treated with 15% dextrose prolotherapy around and inside the knee, 2 times with a two-week interval, and home exercise program (isometric and isotonic exercises).
  Interventions: Drug: Dextrose prolotherapy injection

INTERVENTIONS:
Drug: Dextrose prolotherapy injection — 15% dextrose prolotherapy injection into the knee and 15% dextrose prolotherapy injection will be applied to the painful adhesions of the ligaments around the knee.
  Arms: Dextrose prolotherapy treatment
Combination Product: conventional physical therapy — 4 weeks (20 sessions) physical therapy (Hotpack, TENS and Ultrasound) and home exercise program (isometric and isotonic exercises).
  Arms: Conventional physical therapy

SUMMARY:
Osteoarthritis is a degenerative joint disease characterized by erosion of the articular cartilage, bone hypertrophy at the margins of the joint, subchondral sclerosis, and some biochemical and morphological changes in the synovial membrane and joint capsule. It is the most common joint disease that causes serious morbidity and its prevalence increases with age. It is known that there is a decrease in the muscle strength around the knee in knee osteoarthritis, which creates difficulties in daily living activities.

Prolotherapy is a regenerative treatment method in the treatment of chronic musculoskeletal pain, in which an irritating solution is injected, often hypertonic dextrose, into painful ligament and tendon attachments and adjacent joint spaces.

In this study, it is aimed to investigate the effect of dextrose prolotherapy application in and around the knee on pain, range of motion and knee flexor/extensor muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 50-75 years
* 2-3 knee osteoarthritis by Kellgren Lawrence stage
* Knee pain and functional limitation

Exclusion Criteria:

* Past knee surgery
* Intra articular knee injections in the last six months
* Symptomatic heart and lung disease
* Joint contracture
* History of malignant disease
* Bleeding disorder

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Knee osteoarthritis is more common in women.
Enrollment: 60 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | VAS will be evaluated 3 times before treatment, 1 and 3 months after treatment. Afterwards, the changes between the pre-treatment and 1st month values and the pre-treatment and 3rd month values will be examined.
  10 cm Visual Analogue Scale (0 best, 10 worst pain)
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | WOMAC will be evaluated 3 times before treatment, 1 and 3 months after treatment. Afterwards, the changes between the pre-treatment and 1st month values and the pre-treatment and 3rd month values will be examined.
  A 24-item scale that assesses pain, stiffness, and physical function for knee osteoarthritis. The questions are evaluated by the participants between 0-4 points and the scale takes a value between 0-96 points in total.
Knee isokinetic power | This will be evaluated 3 times before treatment, 1 and 3 months after treatment. Afterwards, the changes between the pre-treatment and 1st month values and the pre-treatment and 3rd month values will be examined.
  Knee flexion and extension strengths will be evaluated with an isokinetic dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Ogut, Dr., Study Director — Mustafa Kemal University
Locations (1):
- Hatay Mustafa Kemal University Faculty of Medicine, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Farpour HR, Fereydooni F. Comparative effectiveness of intra-articular prolotherapy versus peri-articular prolotherapy on pain reduction and improving function in patients with knee osteoarthritis: A randomized clinical trial. Electron Physician. 2017 Nov 25;9(11):5663-5669. doi: 10.19082/5663. eCollection 2017 Nov. PMID 29403602
- [Result] Rabago D, Patterson JJ, Mundt M, Kijowski R, Grettie J, Segal NA, Zgierska A. Dextrose prolotherapy for knee osteoarthritis: a randomized controlled trial. Ann Fam Med. 2013 May-Jun;11(3):229-37. doi: 10.1370/afm.1504. PMID 23690322